CLINICAL TRIAL: NCT05705661
Title: Randomized, This Study Aims To Investigate the Effect of High Frequency Chest Wall Oscillation in Hospitalized Covid-19 Patients.
Brief Title: INFLUENCE OF HIGH FREQUENCY CHEST WALL OSCILLATION IN HOSPITALIZED PATIENTS WITH COVID-19
Acronym: HFCWO IN COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadeel Ibrahim Elsayed Elhannony, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003890
Record Dates: First submitted 2023-01-28; First posted 2023-01-31 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: COVID-19
Keywords: HFCWO; COVID
MeSH Terms: conditions — COVID-19 | interventions — Chest Wall Oscillation

STUDY DESIGN:
Intervention Model Description: A. Subject selection:
  After calculating sample size, sixty hospitalized Covid-19 Patients will be assigned into two equal matched groups randomly:
  Group I (Control): will consist of 30 hospitalized covid-19 patients with (nasal cannula/face mask) who will receive traditional respiratory techniques (breathing ex.) plus their traditional medications.
  Group II (Study): will consist of 30 hospitalized covid-19 patients with (nasal cannula/ face mask) who will receive high frequency chest wall oscillation in addition to breathing exercise techniques plus their traditional medications.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The control group (I) (No Intervention): The control group (I): The participants will follow the traditional pulmonary rehabilitation program including (active cycle of breathing technique, breathing control, deep breathing exercises, huffing). The session duration will be between 30 min twice/day for 15 days as guided by subject fatigue and comfort. (According to Borg scale of dyspnea for monitoring).
- The study group (II) (Active Comparator): The study group (II): The participants will receive active cycle of breathing technique, breathing control, deep breathing exercises (15 min) in addition to (HFCWO); the patient position will be in a semi-recline position, with wrapped vest around the chest. The (HFCWO) protocol included 3-5 cycles, with a pressure range of +10 to +40 IP cmH2O and will be adjusted according to the patient age, number of secretions, tolerance of patients, and chest auscultation every session. The numbers of total sets will be 3-5 with a duration of 15 min, daily, for two sessions / day , time range according to the ability of the patient. (Çelik et al., 2021).
  Interventions: Device: HIGH FREQUENCY CHEST WALL OSCILLATION

INTERVENTIONS:
Device: HIGH FREQUENCY CHEST WALL OSCILLATION — The HFCWO device used a triangular wave form which increases the airflow velocity more than other devices. Therefore, clearing sticky airway mucus and alveolar exudates and maintaining airway patency has become currently the most urgent issue in the ventilatory management of patients with severe COVID-19.
  Other Names: The (HFCWO) (Comfort Cough II, SOUTH KOREA).
  Arms: The study group (II)

SUMMARY:
INFLUENCE OF HIGH FREQUENCY CHEST WALL OSCILLATION IN HOSPITALIZED PATIENTS WITH COVID-19

The purpose of this Interventional study is to investigate the effect of high frequency chest wall oscillation in hospitalized COVID-19 patients on:

1. Inflammatory markers: Netrophil to lymphocyte ratio and CRP
2. Hemodynamic parameters (Arterial Blood Gases, Heart Rate variability, Respiratory Rate, O2 Saturation).
3. Dyspnea, time needed for oxygen weaning, Mortality Rate and Hospital stay period.

Hypotheses :

This Interventional study will test the following Null hypothesis:

* HFCWO will not have an effect in hospitalized COVID-19 patients regarding Arterial Blood Gases, CRP, Dyspnea, Heart Rate variability, Respiratory Rate, O2 Saturation, time needed for Oxygen Weaning, Mortality Rate and Hospital Stay Period.Research Question:
* Is there a significant effect of high frequency chest wall oscillation (HFCWO) in Hospitalized COVID-19 Patients?

DETAILED DESCRIPTION:
Novel coronavirus disease 2019 (COVID-19) infections, declared by the World Health Organization (WHO) as a pandemic, had unprecedented global effects on people's daily activities and way of life.

High-frequency chest wall oscillation (HFCWO) have been shown to be effective at loosening and removing airway mucus in hospitalized people. Mucus weight was greater after HFCWO than after traditional airway clearance interventions involving postural drainage and manual percussion and vibration techniques.

Earlier diagnosis of COVID-19 may be facilitated by heart rate (HR) and heart rate variability (HRV) monitoring. HR and HRV parameters could not only help to detect COVID-19 in a timely manner but could also help to identify patients at risk for cardiovascular/pulmonary complications. Additionally, HRV and HR parameters may help to assess the course of the disease.

The World Health Organization indicates that a resting value of RR > 30 breaths/min is a critical sign for the diagnosis of severe pneumonia in adults, while the cut-off value for children varies according to age.

ELIGIBILITY:
Inclusion Criteria:

1. Sixty hospitalized covid-19 patients from both genders their ages will be ranged from 55 - 65 years old.
2. Desaturated covid-19 patients with lung fibrosis are diagnosed by the physician and confirmed by chest CT
3. Duration of illness ranged from 1 week to 2weeks.
4. All patients have resting oxygen saturation (SpO2) from 80 - 92 %
5. O2 therapy is delivered via Nasal cannula or face mask.
6. All patients will approve and sign a consent form before starting the program which will include the purpose, natures and potential risks of the study which will be explained to all patients (Appendix I).

Exclusion Criteria:

1. Hemodynamically unstable patient
2. Patient with pneumothorax (if chest tube is present)
3. Asthmatic patient
4. Patient with chest deformities
5. Patient with pleural effusion
6. Patient with diaphragmatic hernia
7. Patient with cardiac and thoracic surgery
8. Mechanically Ventilated and intubated patients.
9. Metabolic or cardiovascular diseases.
10. Patients have (SpO2) less than 80 %.
11. Patient with severe lung fibrosis.

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Arterial blood gasses (ABG) | 2 weeks
  Arterial blood gas analysis is a common investigation in emergency departments and intensive care units for monitoring patients with acute respiratory failure. ABG also has some applications in general practice, such as assessing the need for domiciliary oxygen therapy in patients with chronic obstructive pulmonary disease. An arterial blood gas result can help in the assessment of a patient's gas exchange, ventilator control and acid-base balance. (Verma et al., 2010)
Netrophil to lymphocyte ratio | 2 weeks
  The neutrophil-to-lymphocyte ratio (NLR) is an inflammatory marker derived from combining the absolute blood neutrophil and lymphocyte counts, two routinely performed parameters in clinical settings. Recently, studies have reported that NLR levels were higher in more severe patients and were suggested to confer a prognostic value in COVID-19 patients (Lagunas et al.,2020).
heart rate variability | 2 weeks
  Earlier diagnosis of COVID-19 may be facilitated by heart rate (HR) and heart rate variability (HRV) monitoring. HR and HRV parameters could not only help to detect COVID-19 in a timely manner but could also help to identify patients at risk for cardiovascular/pulmonary complications. Additionally, HRV and HR parameters may help to assess the course of the disease. (Buchhorn et al., 2020).
respiratory rate | 2 weeks
  The World Health Organization indicates that a resting value of RR > 30 breaths/min is a critical sign for the diagnosis of severe pneumonia in adults, while the cut-off value for children varies according to age (World Health Organization, 2020).
  Resting RR values also contribute to the prognosis of COVID-19 patients as ICU admission and mortality are associated with significantly higher RR values compared to non-ICU patients and survivors (Huang et al., 2020 & Zhou et al., 2020).
O2 saturation | 2 weeks
  Levels of dyspnea appear to vary significantly amongst patients suffering from COVID-19 ranging from 18.6 to 59%. (Guan et al., 2020). More recently, Li et al (2020) systematic review on 1,994 COVID-19 patients showed an overall percentage of patients experiencing dyspnea was 21.9% in addition. Huang et al. found a prevalence of breathlessness as high as 92% amongst COVID- 19 patients hospitalized in intensive care units versus 37% in non-intensive care units. (Huang et al.,2020).
CRP | 2 weeks
  C-reactive protein) CRP) was an independent risk factor for severe COVID-19. The optimal working point was 38.55 mg/L. This is consistent with previous research showing that hypoalbuminemia, lymphopenia, and CRP more than equal to 40 mg/L were the predictive factors for pneumonia progression to respiratory failure (Ko et al., 2016). Besides, higher CRP has been linked to unfavorable aspects of COVID-19 diseases, such as cardiac injury, and ARDS development, and death. (Terpos et al., 2020).

SECONDARY OUTCOMES:
dyspnea questionnaire | 2 weeks
  The Dyspnea-12 (D-12) Questionnaire is a convenient patient-reported scale for measuring the severity of breathlessness. Breathlessness is quantified by using 12 descriptors to cover both the physical and the psychological dimensions. The D-12 has established its validity and reliability in COPD, asthma, interstitial lung disease, and pulmonary hypertension. (Yorke et al., 2010).
Hospital Stay | one month
  Severe COVID-19 patients were more likely to present with higher levels of inflammation upon hospital admission.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadeel Elhannony, Cairo, Cairo Governorate, Egypt

REFERENCES:
- [Background] Celik M, Yayik AM, Kerget B, Kerget F, Doymus O, Aksakal A, Ozmen S, Aslan MH, Uzun Y. High-Frequency Chest Wall Oscillation in Patients with COVID-19: A Pilot Feasibility Study. Eurasian J Med. 2022 Jun;54(2):150-156. doi: 10.5152/eurasianjmed.2022.21048. PMID 35703523
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143